CLINICAL TRIAL: NCT04483349
Title: "What Do You Value?" A Survey Study Assessing How Patients and Health Care Providers Weigh the Different Components of the Value Equation
Brief Title: Assessment of What Patients and Healthcare Providers Value
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2020-0211; NCI-2020-04577 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0211 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2020-07-14; First posted 2020-07-23 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Gastric Adenocarcinoma; Pancreatic Adenocarcinoma; Pancreatic Neuroendocrine Carcinoma
MeSH Terms: conditions — Somatostatinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (survey administration): Patients and healthcare providers complete a survey over 10-15 minutes.
  Interventions: Other: Survey Administration

INTERVENTIONS:
Other: Survey Administration — Complete survey

SUMMARY:
To assess the importance patients place on each of the attributes of value (i.e., outcomes, quality of life [QOL], cost, experience), and how these patientsâ€™ views differ depending on the stage of their therapy (pretreatment, preoperative therapy, post-operative, long-term surveillance, recurrence).

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the importance patients place on each of the attributes of value (i.e., outcomes, quality of life [QOL], cost, experience).

SECONDARY OBJECTIVES:

I. To assess which attributes of value (i.e., outcomes, QOL, cost, experience) health care providers (i.e., physicians, nurses, administrators) feel are most important in health care delivery.

II. To assess how these patients' views differ depending on the stage of their therapy (pretreatment, preoperative therapy, post-operative, long-term surveillance, recurrence).

III. To assess how patients' view differ to health providers.

OUTLINE:

Patients and healthcare providers complete a survey over 10-15 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Any patient who has been treated, or is anticipated to be treated, for potentially resectable, biopsy-proven pancreatic adenocarcinoma, pancreatic neuroendocrine malignancy, or gastric adenocarcinoma
* Providers involved in the care of gastric and pancreatic cancer patients. Providers will include non-collaborative surgical oncologists, medical oncologists, radiation oncologists, administrators, nurses, mid-level providers
* Able to understand the description of the study and willing to participate

Exclusion Criteria:

* Inability to read and answer questions in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pancreatic adenocarcinoma, pancreatic neuroendocrine malignancy, or gastric adenocarcinoma, and healthcare providers involved in the care of gastric and pancreatic cancer patients at the MD Anderson Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 397 (Actual)
Dates: Start 2020-06-11 (Actual); Primary Completion 2022-08-11 (Actual); Study Completion 2022-08-11 (Actual)

PRIMARY OUTCOMES:
Importance patients place on each of the attributes of value (i.e., outcomes, quality of life [QOL], cost, experience) | Survey completion up to 1 year
  We will calculate the mean rank of patients yielding usable data and its corresponding 95% confidence interval. Patient characteristics and survey items will be summarized using descriptive statistics, including means, standard deviations (SDs), proportions, range, and 95% confidence intervals (CIs), etc.

SECONDARY OUTCOMES:
Most important attributes of value to healthcare providers | Survey completion up to 1 year
  Provider characteristics and survey items will be summarized using descriptive statistics, including means, SDs, proportions, range, and 95% CIs, etc.
Importance care providers (i.e., physicians, nurses, administrators) place on each of the attributes of value (i.e., outcomes, quality of life [QOL], cost, experience) | Survey completion up to 1 year
  Chi-square tests (or Fisher's exact test) will be used to compare the results between patients and providers.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew H Katz, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: Related Info — http://www.mdanderson.org